CLINICAL TRIAL: NCT06880510
Title: The Locus Coeruleus, Norepinephrine and Cognitive Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1910009087
Record Dates: First submitted 2024-03-22; First posted 2025-03-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cornell University (Experimental): Short-duration (less than an hour) vagus nerve stimulation will be delivered while participants engage in cognitive tasks and games. This study also includes a 90-minute MRI, blood pressure testing, saliva collection for genetic analysis, sensory testing, and blood pressure/heart rate measurement.
  Interventions: Device: t-VNS transcutaneous auricular vagus nerve stimulator

INTERVENTIONS:
Device: t-VNS transcutaneous auricular vagus nerve stimulator — An investigator will clip the the transcutaneous auricular vagus nerve stimulator (taVNS) to the outer ear, and apply electrical current to modulate the activity of the vagus nerve. During this process, the investigator will monitor pupil size and heart rate to determine whether either of these variables is affected by vagus nerve stimulation.

SUMMARY:
The locus coeruleus (LC) has recently been identified as one of the earliest sites of damage in AD with pathological lesions appearing as early as the mid-20s. In this study, the investigators use a variety of techniques including structural MRI, functional MRI, pupillometry, and transcutaneous vagus nerve stimulation to assess the health of the LC and its relation to easily measurable peripheral variables.

DETAILED DESCRIPTION:
Unfortunately, most people are personally familiar with the devastating consequences of neurodegenerative disorders such as Alzheimer's disease (AD) and Parkinson's disease (PD). The number of older adults with neurodegenerative disease is expected to rise as the baby boomer generation ages, with 28 million baby boomers developing AD. This, in turn, is expected to cost $328 billion dollars, or 24% of total Medicare spending. Despite decades of research into the causes of AD, there are only 5 FDA-approved treatments, all of which are supportive, non-disease-modifying drugs. Of the treatments that have been tested for AD, 99.6% have failed. Accordingly, new approaches to neurodegenerative disease - a better understanding of their causes and better targets for treatment - are desperately needed.

The locus coeruleus (LC) has recently been identified as one of the earliest sites of damage in AD and PD, with pathological lesions appearing as early as the mid-20s. A brain region of 40,000-60,000 neurons located in the brainstem, the LC is the source of the neurochemical norepinephrine (NE, also known as noradrenaline). The LC has widespread projections throughout the nervous system and plays an important role in arousal, attention, memory, mediation of emotional and stress responses, and some aspects of motor control. Damage to the LC, and the resulting decrease in protective NE signaling throughout the brain, is proposed to be an important mechanism in the progression of neurodegeneration. The LC has even been proposed by some to be the primary mediator of cognitive reserve, predicting the relative preservation of cognitive performance despite neuropathological insult. Despite the possibility that decreased NE signaling from the LC may serve as the earliest warning flag of dementia, few studies link LC function and cognitive performance. Remarkably, neither has the relationship between LC function and LC neuronal loss been examined. A promising new technique, neuromelanin-sensitive magnetic resonance imaging (MRI), will allow us to estimate the amount of neuromelanin-containing tissue in the LC. Neuromelanin MRI has been shown to be quantitative, highly correlated with the number of LC neurons, and reproducible, with high inter-rater reliability. The investigators have been using this innovative technique to establish a correlation between LC neuromelanin density and attention across the lifespan, which may provide a non-invasive, functional measure of neurodegeneration risk that may be valid well before the onset of clinical symptoms. Furthermore, using modern MRI analysis techniques, it is now possible to measure the function of the LC with functional MRI.

As an even less invasive measure of LC function, the investigators propose to assess task-evoked pupillary responses during auditory and visual vigilance tasks. Light-evoked pupillary responses - changes in pupil size due to changes in illumination - are well known to be abnormal in AD, but task-evoked pupillary responses may represent an early sign of future cognitive decline. Pupil diameter, under constant light conditions, is a well-established correlate of neuronal activity in LC neurons. Measuring pupil changes with a non-invasive eyetracker is an ideal assay for this purpose.

To further characterize the relationship between LC integrity, LC function, and cognitive function the investigators will administer a broad neuropsychological battery to measure cognitive performance. The laboratory makes use of a variety of classic neuropsychological tests such as the Montreal Cognitive Assessment and Trail-Making Test, in addition to the NIH Toolbox Cognition and Emotion Batteries, blood pressure and other cardiovascular health measurements, a retrospective report of traumatic childhood experiences, and a variety of custom-designed attention tasks for use with the MRI scanner and eyetracking components of the study.

There is intriguing neurogenetic evidence that individual differences in NE signaling may protect against AD. A common polymorphism (small genetic change) in the adrenergic receptor alpha 2b gene (a molecule in the brain that binds to norepinephrine, "adra2b deletion variant") likely results in significantly increased NE signaling from the LC. The lab has previously shown that individuals with this polymorphism attend to and later recall emotional events better than those without, and experience greater perceptual vividness. Crucially - others have shown that individuals with this polymorphism are less likely to have AD or mild cognitive impairment. These phenomena are likely all related to the role that the LC plays in attention, arousal and, in combination, support healthy cognitive aging.

Finally, the investigators will also attempt to modulate LC activity using non-invasive transcutaneous auricular vagus nerve stimulation for very short periods (~15 to 45 minutes) to discover if it is possible to alter, and potentially improve, LC function variables. Previously, this technique has been shown to directly activate the LC through the vagus nerve.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Able to speak and understand English
* Hearing and vision correctable to normal or near-normal
* Willing and able to use a touchscreen
* Willing and able to use a keyboard and mouse
* Willing and able to undergo a MRI scan at the Cornell MRI Facility lasting approximately 90 minutes.

Exclusion Criteria:

* Moderate or severe brain injury
* Serious neurological disorders such as epilepsy
* Recent concussion
* Colorblindness
* Use of street drugs
* Cardiac arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Tonic pupil size in mm | 15-45 minutes
  The investigators will continuously monitor tonic pupillary size to determine whether it is affected by taVNS. To do so, the investigators will use a EyeLink 1000+ eyetracker and measure pupil diameter continuously throughout the completion of computer-based cognitive tasks, such as an Oddball task, Attentional Boost Effect task, Proactive Interference task, or Tone Gap task. Tonic pupil size are measured with custom software, and pupil size is reported in mm.
Heart rate variability | 15-45 minutes
  The investigators will continuously monitor heart rate using photoplethysmography (BIOPAC Systems) to calculate heart rate variability, to determine whether it is affected by taVNS. Root mean square of successive differences (RMSSD) will be the specific heart rate metric used.
Discriminability index on tests including the attentional boost effect task | 15-45 minutes
  The investigators will test performance on measures of attention (e.g. Oddball paradigm, Flanker inhibitory control paradigm, attentional boost effect paradigm) to determine whether performance on this task, specifically d' (discriminability index) is affected by taVNS.
Phasic pupillary responses in mm | 15-45 minutes
  The investigators will monitor phasic pupillary response size to determine whether they are affected by taVNS. To do so, the investigators will use a EyeLink 1000+ eyetracker and measure pupil diameter continuously throughout the completion of computer-based cognitive tasks, such as an Oddball task, Attentional Boost Effect task, Proactive Interference task, or Tone Gap task. Phasic pupil sizes are measured with custom software, and response size is reported in mm.
Reaction time on tests including the attentional boost effect task | 15-45 minutes
  The investigators will test performance on measures of attention (e.g. Oddball paradigm, Flanker inhibitory control paradigm, attentional boost effect paradigm) to determine whether performance on this task, specifically reaction time, is affected by taVNS.

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Completely de-identified participant data (with no demographic data that could reasonably result in identification) may be given to other researchers on request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Indefinitely.
Access Criteria: The data may be posted on Open Science Framework if required by publications.
URL: https://osf.io/